CLINICAL TRIAL: NCT06897878
Title: OPTImal Number of Pleural BIOPsies During Pleuroscopy
Acronym: OPTIBIOP
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Udit Chaddha, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-24-01325
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Pleural Diseases
Keywords: Pleuroscopy; Pleural effusion; Pleural biopsy
MeSH Terms: conditions — Pleural Diseases; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pleural tissues from pleural biopsies that will be analyzed in the pathology lab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pleural biopsy: All consecutive patients referred for a pleuroscopy.

SUMMARY:
A single-center, non-randomized, prospective observational, pilot study designed to determine what is the optimal number of pleural biopsies to take during pleuroscopy.

DETAILED DESCRIPTION:
After enrollment, participants will undergo pleural biopsies via pleuroscopy. Specimens will be divided into three aliquots (1-3, 4-6, 7-10), which will be sent to pathology. A designated pathologist will evaluate the specimens in each aliquot to determine the number of biopsies required to reach a diagnosis and to obtain sufficient material for biomarker testing (when needed), and determine whether analysis of further aliquots is needed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients who require pleuroscopies will be enrolled to the study.
* Age ≥ 18

Exclusion Criteria:

- Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients that undergo pleuroscopy for pleural biopsies, excluding those with inability to provide informed consent.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Number of pleural biopsies to reach a diagnosis | At week 2 after pleuroscopy
  The number of pleural biopsies needed to reach a diagnosis.

SECONDARY OUTCOMES:
Number of pleural biopsies required for comprehensive biomarker testing. | At week 4 after pleuroscopy
  The number of biopsies required to obtain sufficient material for comprehensive biomarker testing.
Number of complications | At week 4 after pleuroscopy
  Number of complications related to the biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Udit Chaddha, Principal Investigator — MBBS
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data. Any purpose. Proposals should be directed to jeeyune.bahk@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.